CLINICAL TRIAL: NCT02430883
Title: Is There Any Relation Between Pain and Stone Location in Retrograde Intrarenal Surgery?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Nihat Karakoyunlu, MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 15.12.2014 18/15
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Nephrolithiasis
Keywords: pain, RIRS, kidney
MeSH Terms: conditions — Nephrolithiasis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- first group (Active Comparator): patients who have upper pole kidney stones treated with flexible renoscopy
  Interventions: Procedure: Retrograde Intrarenal Surgery
- second group (Active Comparator): patients u who have mid pole kidney stones treated with flexible renoscopy
  Interventions: Procedure: Retrograde Intrarenal Surgery
- third group (Active Comparator): patients who have lower pole kidney stones treated with flexible renoscopy
  Interventions: Procedure: Retrograde Intrarenal Surgery
- forth group (Active Comparator): patients who have kidney stones in pelvis treated with flexible renoscopy
  Interventions: Procedure: Retrograde Intrarenal Surgery
- fifth group (Active Comparator): patients who have multiple calixes kidney stones treated with flexible renoscopy
  Interventions: Procedure: Retrograde Intrarenal Surgery

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery — endoscopic treatment of kidney stones with flexible renoscopy

SUMMARY:
We want to serach the relationship between the pain degree and stone localisation in kidney in Retrograde intrarenal surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing RIRS Age between 18 and 90 years

Exclusion Criteria:

* Patients who have congenital urogenital abnormalities 2)Patients who have previous surgery history

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Pain degree | Pain degree postoperative 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dıskapı TRH, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Polito C, La Manna A, Signoriello G, Marte A. Recurrent abdominal pain in childhood urolithiasis. Pediatrics. 2009 Dec;124(6):e1088-94. doi: 10.1542/peds.2009-0825. Epub 2009 Nov 9. PMID 19901004